CLINICAL TRIAL: NCT06192381
Title: Effect of Applying Web-Based Health Education Module on Nursing Students' Knowledge, Adaptive Healthy Measures and Attitude Regarding Polycystic Ovary Syndrome: A Randomized Controlled Trial
Brief Title: Effect of Web-Based Module on Nursing Students' Knowledge, Practice and Attitude Regarding Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Safa Hamdy Alkalash Alsayed (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor-Investigator, Safa Hamdy Alkalash Alsayed, Assistant professor of family medicine, Umm Al-Qura University
Organization: Umm Al-Qura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: No.P.0360
Record Dates: First submitted 2023-11-28; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: PCOS
Keywords: Web-Based Learning Model; Knowledge; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: A two-armed, single-blind, parallel groups prospective randomized controlled trial (RCT), with a baseline pre-test and immediate post-test was used to carry out this study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional health education group (control group) (No Intervention): Traditional health education group (control group) (n = 68) who received health education with the traditional face-to-face method
- web-based health education group (intervention group) (Experimental): Web-based health education group (intervention group) (n = 68) who received health education with the Web-Based Learning Module (WBL).
  Interventions: Other: Web-Based Learning Module (WBL)

INTERVENTIONS:
Other: Web-Based Learning Module (WBL) — To ensure a uniform starting point, the participants were recruited via faculty website and students' academic counseling services. At the baseline, after the initial assessment, the participants were randomized at a 1:1 allocation ratio into the following groups: 1) traditional health education group (control group) (n = 68) who received health education with traditional face-to-face method; 2) web-based health education group (intervention group) (n = 68) who received health education with Web-Based Learning Module (WBL).
  Arms: web-based health education group (intervention group)

SUMMARY:
Background: Polycystic ovary syndrome (PCOS) is a heterogeneous endocrinopathy among reproductive-aged women that has become a major international public health concern. Objective: Investigate the effect of web-based health education module on nursing students' knowledge, adaptive healthy measures and attitude regarding polycystic ovary syndrome. Research design: A two-armed, single-blind, parallel groups prospective randomized controlled trial (RCT), with a baseline pre-test and immediate post-test was used to carry out this study. Setting: The study was conducted at the Faculty of Nursing, Mansoura University, Egypt in December 2022 to May 2023. Subjects and sampling: Simple random sampling technique was employed to recruit the study subjects. Data collection: A questionnaire was developed to acquire data including six parts.

DETAILED DESCRIPTION:
Pre-intervention phase:

Initial data was gathered about the participants' socio-demographic characteristics, their knowledge, adaptive healthy measures, and attitude toward PCOS before the implementation of the health education intervention. A brief introduction to the goals, processes, voluntary nature of participation, confidentiality and anonymity declarations, and questionnaire cover page were all included. Participants were made aware that they could withdraw from the study at any moment, there would be no negative repercussions, and they could choose to have any case data acquired for the study destroyed. The informed consent form must be signed by the participants and submitted back by ordinary mail to participate.

The developed health education module was created based on the participants' preliminary assessment results and according to recommendations from [30]. It consisted of seven interactive modules (4 hours' sessions) in Arabic that covered the following topics: "overview of PCOS, etiology and risk factors, signs and symptoms, diagnosis, complications, preventive measures, and treatment of PCOS." It aimed at increasing health awareness regarding PCOS, encouraging and promoting adaptive healthy measures to prevent PCOS, and promoting a positive attitude regarding PCOS.

The module development team gathered to discuss how each module would be prepared and formatted, as well as how the modules' sessions would be broken down. The program was designed with a defined purpose, precise goals, pertinent materials, and instructional techniques. In addition, it was developed to provide easy access to web-based education that incorporates sources to increase knowledge and support healthy measures and a positive attitude regarding PCOS. This is done using a set of technical and instructional standards developed by a web-based design team and an information technology expert. The researchers provided the web designer with word-processed documents representing each distinct learning session, videos, a storyboard of suggested graphics, and a description of interactions.

The development team met once a week to go over any issues that might occur with the module, to offer ideas and comments where appropriate, and to address any queries that might have come up while each session was being developed. The web-based design team and researchers chose a learning platform that gave users access to data, tools, and resources to support the administration and delivery of education about PCOS and associated preventive actions online. To get rid of Wix's pop-up advertisements, the researchers bought a distinctive website domain URL.

The site map and links to the tutorials, forums, and other resources are all accessible from the main screen. The web-based module also included a chat room where students and students conducting research could post questions and engage in conversation. To get user feedback on the learning experience and improve the interface, post-learning discussions and comments were created. Additionally, each student's frequency and amount of time spent were noted.

To make it simple for the user to choose another menu, the primary menu is also continuously shown on the upper bar. No session could be skipped because the navigation was sequential from session 1 to session 7. The intervention group participants could move on to the following screen, replay the current screen, or go back to the previous screen at any time during a session. They were given as much time as they needed to consider the data displayed on each screen.

The researchers developed the content of the web-based health education sessions. Besides, they drew lines between the elements to indicate how they were linked together. These lines helped dictate sessions' organization, navigation, and hyperlinks. Moreover, it was arranged into seven sessions. It was displayed by using text, pictures, and videos.

The content was uploaded to the website by the researchers and professional programmers (https://healthconcerns.tech/). The link to the website was distributed to a panel of five external reviewers (experts in community health nursing, women's health and midwifery nursing, and professional programmers) to systematically test the content's validity, clarity, consistency, accuracy, applicability, and format before the application of the web-based education module. Any specific guidelines or suggestions from the experts' evaluation were recorded and considered while creating the web-based teaching sessions. The traditional training session that was given to the control group's students' material was the same.

The face validity of the web-based modules was assessed concurrently with the review process using a sample group of students (n = 14) who had no prior knowledge of PCOS to assess the clarity, applicability, and reliability of the module and to determine the approximate time needed to implement these sessions. Each student in the intervention group completed a module each week and gave the content producer detailed comments afterward. In most cases, students' input noted areas that needed clarification and more examples, as well as those that were unclear and confusing. During the revision process, student feedback was considered. By clicking on the link, participants could view the questions and submit their responses.

Intervention phase:

The intervention condition: The research website was recommended to the students in the intervention group of the study who had completed the pre-self-administered questionnaires. There, they learned more about the study and what participating in it entailed. The members of the intervention group were forced to create accounts on the website using personal passwords after logging in. An informational session was conducted to teach the intervention group's members how to utilize the learning management system (LMS) before they started their virtual education. The participants were given instructions to complete the module on their own for the duration of the session after receiving a brief orientation to the navigational features in addition to the help screen in the module. The module can be used on mobile devices, laptops, and personal computers. The online education module was only given to the intervention group.

The intervention group's participants were permitted to access the module as many times as necessary to finish all of the sessions (https://healthconcerns.tech/). The participants were instructed to finish at least one and no more than two modules per week. Each module took 30 to 60 minutes to complete. The intervention was therefore planned to be finished in roughly 5 to 7 weeks. They were also told to heed the health advice that was given. Through website chat, all of the participants' inquiries were addressed, and they received feedback.

The control condition is: Regarding the traditional health education group, the students had full access to traditional face-to-face health education regarding PCOS for a similar duration and by the same researchers. They were divided into seven groups. Each group had nine to ten students. The nursing faculty's instructional hall served as the location for the sessions. Each group's session lasted 5 hours over 2 days per week (10 a.m.-12 p.m.). Lectures, discussions, brainstorming, blackboards, printed handouts, and audiovisual materials were employed as teaching and learning tools throughout the sessions.

post-intervention phase Participants' knowledge, adaptive healthy measures, and attitude about PCOS were evaluated using the same pre-test questionnaire for the intervention group and the control group. Additionally, feedback about the website was assessed once after completion of the module for the intervention group. All participants from the intervention and control groups started and completed the PCOS educational module. The control group was invited and given access to receive the identical web-based instructional module once data collection, evaluation, and analysis were finished.

ELIGIBILITY:
Inclusion Criteria:

The target population of this study was nursing students at all academic levels enrolled in a bachelor-level in the Faculty of Nursing. The following inclusion requirements (female university undergraduate nursing students, had no significant co-morbidity and declared willingness to provide self-report data at the two assessment points). For the intervention group, familiarity with and internet access should be emphasized.

Exclusion Criteria:

Exclusion criteria were (nursing students with PCOS who were already receiving treatment, and non-consenting participants).

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2022-12-11 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
The primary outcomes were improvement of students' knowledge, adaptive healthy measures and attitude regarding PCOS | 12 months
  The primary outcomes were improvement of students' knowledge, adaptive healthy measures and attitude regarding PCOS. The primary outcomes was measured using the study questionnaire (Parts: 3-4 & 5) pre and post-intervention.

SECONDARY OUTCOMES:
The secondary outcome was students' satisfaction with the web-based educational sessions. | 12 months
  The secondary outcome was students' satisfaction with the web-based educational sessions. The secondary outcome was measured using the study questionnaire (Part: 6), once post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Safa H Alkalash, MD, Principal Investigator — Umm Al-Qura Univeristy
Locations (1):
- Faculty of Nursing, Mansoura University,, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamed RA, Taref NN, Osman NE, Keshta NHA, Alboghdady MA, Marzouk MM, Almowafy AA, Fadel EA. Effect of web-based health education on nursing students' knowledge, adaptive healthy measures and attitudes regarding polycystic ovary syndrome: a randomized controlled trial. BMC Nurs. 2024 Jul 15;23(1):479. doi: 10.1186/s12912-024-02015-7. PMID 39010089